CLINICAL TRIAL: NCT03773276
Title: Norepinephrine Boluses for Prevention of Postreperfusion Syndrome in Living Donor Liver Transplantation
Brief Title: Norepinephrine Boluses in Liver Transplantation
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R.18.11.323 - 2018/11/05
Record Dates: First submitted 2018-12-03; First posted 2018-12-12 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Living Donor Liver Transplantation; Norepinephrine Bolus; Postperfusion Syndrome

STUDY DESIGN:
Intervention Model Description: This is a feasibility (efficacy and safety) trial that tests the Norepinephrine boluses for the prevention of postreperfusion syndrome during liver transplantation operation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Norepinephrine boluses (Experimental): Single arm study
  Interventions: Drug: Norepinephrine boluses

INTERVENTIONS:
Drug: Norepinephrine boluses — On portal vein declamping, We will inject NE boluses in the C.V.P port of the pulmonary artery catheter with 5 ml saline flushing after each. After reperfusion, we will start bolus noradrenaline 20 µg if mean arterial blood pressure (mABP) decreases by 10 % or more of the basal reading (immediately before portal vein declamping after ensuring withholding of the surgical manipulation). Additional NE boluses will be given as follow;
  * If mABP rises to 65 mmHg (lowest target level), we will hold NE boluses.
  * If mABP remains constant or begins to rise but did not reach 65 mmHg, we will give 20 µg after 10 seconds from the previous bolus
  * If mABP continues to drop, we will add 10 µg to the previous dose after 10 seconds and can be repeated.
  * If mABP remains below 65 mmHg more than 1 minute, we will give the scheduled bolus NE with adding 10 µg adrenaline boluses.
  Other Names: Noradrenaline boluses

SUMMARY:
We study the efficacy of Norepinephrine boluses on prevention of postreperfusion syndrome during living donor liver transplantation.

NE and Post-reperfusion:

On portal vein declamping, we will start rapid 500 ml 4% albumin infusion or packed RBCs (according to the anhepatic hemoglobin level 5 min before declamping) through 14 Gauge peripheral venous cannula in all patients.

NE boluses technique; We will inject NE boluses in the C.V.P port of the pulmonary artery catheter with 5 ml saline flushing after each. After reperfusion, we will start bolus noradrenaline 20 µg if mean arterial blood pressure (mABP) decreases by 10 % or more of the basal reading (immediately before portal vein declamping after ensuring withholding of the surgical manipulation). Additional NE boluses will be given as follow;

* If mABP rises to 65 mmHg (lowest target level), we will hold NE boluses.
* If mABP remains constant or begins to rise but did not reach 65 mmHg, we will give 20 µg after 10 seconds from the previous bolus
* If mABP continues to drop, we will add 10 µg to the previous dose after 10 seconds and can be repeated.
* If mABP remains below 65 mmHg more than 1 minute, we will give the scheduled bolus NE with adding 10 µg adrenaline boluses.

DETAILED DESCRIPTION:
Anesthesia technique:

On admission to the pre-anesthetic room, patients will receive intravenous pantoprazole sodium 40 mg, midazolam 0.02 mg/kg and the prophylactic antibiotics.

In the operating room, we apply standard monitors in the form of pulse oximetry, non-invasive blood pressure, and electrocardiography. Induction of anesthesia will be fentanyl 2 µg/kg, propofol 1-2 mg/kg, and rocuronium bromide 0.8 -1 mg/kg.

After tracheal intubation, we will insert an arterial catheter in the radial artery of the non-dominant hand after performing modified Allen's test. Then, we will insert five port pulmonary artery catheter for continuous cardiac output monitoring (the equipment).

Anesthesia will be maintained by sevoflurane in 40% oxygen with infusion of fentanyl 0.5-1 µg/kg/h and rocuronium bromide 200-400 µg /kg/h. We adopt goal directed fluid replacement protocol keeping the target mABP of 65 mmHg using norepinephrine in fluid non-responders with low SVR (German medical association 2009). Crystalloids will be Ringer's Acetate and the colloid will be albumin 4% in Ringer Acetate solution.

We will keep the intraoperative and the two-day postoperative glucose between 110 and 180 mg/dl by intravenous insulin infusion or glucose 10% or 25% boluses as appropriate. We monitor UO hourly in the intraoperative and ICU periods and only administer frusemide to prevent volume overload.

Surgical technique:

The donor surgical team will excise the right liver lobe (without inclusion of the middle hepatic vein). They will flush the graft with 3-4 liters of cold histidine-tryptophan-ketoglutarate (HTK) (Custodial, Bensheim, Germany) via antegrade flushing of the portal vein to get completely clear fluid without flushing via the hepatic artery. Both recipient and donor operations will be synchronized to minimize graft preservation time.

The right hepatic vein will be unclamped then the portal vein and the graft preservative contents will be washed into the systemic circulation by the portal blood.

NE and Post-reperfusion:

On portal vein declamping, we will start rapid 500 ml 4% albumin infusion or packed RBCs (according to the anhepatic hemoglobin level 5 min before declamping) through 14 Gauge peripheral venous cannula in all patients.

NE boluses technique; We will inject NE boluses in the C.V.P port of the pulmonary artery catheter with 5 ml saline flushing after each. After reperfusion, we will start bolus noradrenaline 20 µg if mean arterial blood pressure (mABP) decreases by 10 % or more of the basal reading (immediately before portal vein declamping after ensuring withholding of the surgical manipulation). Additional NE boluses will be given as follow;

* If mABP rises to 65 mmHg (lowest target level), we will hold NE boluses.
* If mABP remains constant or begins to rise but did not reach 65 mmHg, we will give 20 µg after 10 seconds from the previous bolus
* If mABP continues to drop, we will add 10 µg to the previous dose after 10 seconds and can be repeated.
* If mABP remains below 65 mmHg more than 1 minute, we will give the scheduled bolus NE with adding 20 µg adrenaline boluses.

Immunosuppression:

All patients will receive intravenous 0.5 gm methylprednisolone at the start of the warm ischemia. After hepatic artery anastomosis and declamping, we will administer 500 mg mycophenolate mofetil through the nasogastric tube and i.v. 20 mg basiliximab.

In the ICU, patients will receive oral tacrolimus starting the day after the operation (adjusting the dose targeting serum level of 5-10 ng/ml) and mycophenolate mofetil 500 mg 4 days after.

In the ICU:

We adopt early ICU tracheal extubation once the patient is hemodynamically stable and pH > 7.3 with adequate consciousness and muscle power (guided by neuromuscular monitoring).

We will keep the pulmonary artery catheter in place for hemodynamic monitoring in case of instability and will exchange it by central venous catheter after 48 hours postoperatively.

Data collection and Monitoring:

1- Preoperative data:

1. Age, sex, weight, height, BSA, MELD score and Child-Pugh classification
2. Medical co-morbidities: hypertension, cardiac diseases, Diabetes Mellitus
3. Cause of the end stage liver disease (ESLD), and the donor age and gender
4. Liver tests: serum albumin, bilirubin, INR, AST, ALT
5. S.Cr
6. C-reactive protein We will collect the preoperative data 24 hours before the operation.

2- Intra-operative and Post-operative data: The primary outcome will be the incidence of PRS. We will record the lowest mABP, the duration of hypotension (below 20% from the basal value or below 65 mmHg). We will record significant arrhythmias, ischemia (ST depression more than 1mV in lead II) during reperfusion and NE boluses. We will report the need and duration of pre-reperfusion and post-reperfusion NE infusions.

We will record the intraoperative CI, SVI, mABP, mPAP, PAOP, SVR, PVR, and serum Na, K, ionized Ca and Cl at six times;

* immediately before skin incision,
* at the beginning of the anhepatic (portal vein clamping),
* 5 minutes before portal reperfusion,
* 5 min after portal unclamping,
* 5 min after hepatic arterial declamping and
* at the time of skin closure. The incidence of the AKI defined as 50% increase in the S.Cr or 0.3 mg/dl increase from the baseline S.Cr in the early 48 post¬operative hours. In the postoperative period, S.Cr will be measured at arrival to ICU, 1st, 2nd, 7th, 28th and at three-month postoperative with measuring of the 24 hour-urine output in the first 2 days.

We will stage AKI as follow: stage 1 when S.Cr = 1.5-1.9 times baseline or > 0.3 mg/dl increase from the baseline, stage 2 when S.Cr = 2-2.9 times baseline and stage 3 when S.Cr = 3 times baseline or increase to > 4 mg/dl or initiation of renal replacement therapy.

We will record warm ischemia, cold ischemia, the total ischemia and the operative times. We will mention the blood transfusions (before and after reperfusion), UO in the anhepatic phase and the total intraoperative amounts.

Laboratory assessment of the graft function will include pH, serum lactate, INR, AST, ALT, GGT, albumin and bilirubin at the 1st, 2nd and 7th days postoperatively. We will report early postoperative surgical complications (7 days) especially vascular insufficiency of the graft detected by the ultrasound Doppler evaluation.

In case of persistent graft dysfunction, graft rejection and ischemia- reperfusion injury will be diagnosed and graded by histopathological examination of liver biopsy performed by consultant liver pathologist.

ELIGIBILITY:
Inclusion Criteria:

* All patients subjected to living donor liver transplantation with right lobe liver graft.

Exclusion Criteria:

1. Acute fulminant hepatitis
2. Chronic hypertension
3. Moderate to severe valvular heart disease
4. Chronic kidney disease (CKD) and Hepatorenal syndrome (HRS)
5. Preoperative S.Cr elevation > 1.4 mg/kg or dialysis recently before surgery
6. Long standing diabetes mellitus (> 10 years on insulin)
7. Moderate and sever Porto-pulmonary hypertension
8. Moderate and sever Hepato-pulmonary syndrome (HPS)
9. Contraindications to pulmonary artery catheter insertion
10. Budd Chiari syndrome
11. Re-transplantation
12. Massive blood transfusion (more than 5 units of blood before portal clamping)
13. Graft/weight ratio > 1.4 and < 0.8

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2020-04-18 (Actual); Study Completion 2020-08-28 (Actual)

PRIMARY OUTCOMES:
Incidence of postreperfusion syndrome | 5 minutes after reperfusion
  PRS defined as 30% drop in the mABP when compared to the mABP just before portal declamping sustained for 1 min within the first 5 min after portal unclamping

SECONDARY OUTCOMES:
Arrhythmia | During and 5 minutes after norepinephrine boluses
  if significant and persistent (or needed treatment or intervention)
Ischemia | During and 5 minutes after norepinephrine boluses
  ST depression more than 1mV in lead II
Liver graft function | After 2 days postoperative
  By pH, serum lactate mmol/l, INR, AST u/ml, ALT u/ml, albumin gm/dl and bilirubin ml/dl as a composite outcome
Acute kidney injury | within the first 2 days postoperative
  50% increase in the S.Cr or 0.3 mg/dl increase from the baseline S.Cr in the early 48 post¬operative hours
3-month survival | 90 days after surgery
  survival within 3 months after liver transplantation
one-year survival | one year after transplantation
  survival for one year post-transplantation as a dichotomous outcome

CONTACTS AND LOCATIONS:
Overall Officials: Amr M Yassen, Professor, Study Director — Mansoura University
Locations (1):
- Mansoura University, Gastrointestinal Surgery Center, Liver Transplantation, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
We will make anonymized individual data available to researchers at appropriate requests. We may make them available as a supplement along with the published manuscript if the journal supports this option.